CLINICAL TRIAL: NCT02542111
Title: A Phase II Study of the Efficacy and Safety of Bortezomib Plus GDP in the Treatment of Refractory and Relapsed Non-GCB Diffuse Large B-cell Lymphoma
Brief Title: A Study of Bortezomib Plus GDP in the Treatment of Refractory and Relapsed Non-GCB DLBCL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, Professor, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: V-GDP
Record Dates: First submitted 2015-08-24; First posted 2015-09-04 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Diffuse Large B-cell Lymphoma
Keywords: diffuse large b-cell lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Bortezomib; Gemcitabine; Dexamethasone; Cisplatin

ARMS (1):
- V-GDP (Experimental): Bortezomib 1.6 mg/m2/d iv d1 and d8 Gemcitabine 1000mg/m2/d iv d1 and d8 Dexamethasone 40mg/d iv d1-4 cisplatin 25 mg/m2 iv d2-4 Frequency every 28 days Total cycles 4
  Interventions: Drug: Bortezomib; Drug: Gemcitabine; Drug: Dexamethasone; Drug: Cisplatin

INTERVENTIONS:
Drug: Bortezomib — Bortezomib IV
Drug: Gemcitabine — Gemcitabine IV
Drug: Dexamethasone — Dexamethasone IV
Drug: Cisplatin — Cisplatin IV

SUMMARY:
This study is to evaluate the efficacy and safety of Bortezomib plus GDP in the treatment of non-GCB DLBCL patients.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven diffuse large B-cell lymphoma non-GCB subtype. Previously treated with 1, and only 1, chemotherapy regimen including an anthracycline and excluding cisplatin, cytarabine, bortezomib and gemcitabine. Relapse after CR, less than PR or PR to previous treatment.
2. No history of stem cell transplantation, and no intention for stem cell transplantation.
3. Age between 16-75.
4. ECOG<3.
5. At least 1 measurable tumor mass.
6. Minimum life expectancy of 3 months.
7. Written informed consent.
8. No uncontrolled CNS involvement by lymphoma:No CNS disease at time of relapse;CNS disease diagnosed at initial presentation allowed provided a complete response for CNS disease was achieved and maintained.

Exclusion Criteria:

1. Chemotherapy or large field radiotherapy within 3 weeks prior to entering the study.
2. Clinically significant active infection.
3. Impaired liver, renal or other organ function not caused by lymphoma, which will interfere with the treatment schedule.
4. Any significant medical or psychiatric condition that might prevent the patient from complying with all study procedures.
5. Subject has ≥grade 2 peripheral neuropathy or grade 1 with pain within 14 days before enrollment.
6. Patients who are pregnant or breast-feeding.
7. HIV infection.

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-05; Primary Completion 2018-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Response rate | Every 2 cycles during treatment and then every 3 months for 2 years
  28 days as one cycle

SECONDARY OUTCOMES:
Progression free survival | 1 year
Overall survival | 1 year
Safety as assessed using the CTCAE | Days 1 of each course and 4-6 weeks after final treatment
  28 days as one cycle

CONTACTS AND LOCATIONS:
Overall Officials: Weili Zhao, Prof, Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China